CLINICAL TRIAL: NCT03509597
Title: A Randomized, Open-Label, Parallel-Group Study to Investigate The Effect of Cognitive Training and Aerobic Exercise on Brain, Functional Outcome and Cognition in Schizophrenia
Brief Title: Brain Image Markers Associated With Cognitive Training and Aerobic Exercise in Schizophrenia
Acronym: CORTEX-SP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Red Salud Mental Araba (Other Government)
Collaborators: University of Deusto (Other); University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CORTEX-SP Study; PI16/01022 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII))
Record Dates: First submitted 2018-04-11; First posted 2018-04-26 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia
Keywords: Cognitive remediation; Aerobic exercise; Physical exercise; Negative symptoms; Functional outcome; Cognition
MeSH Terms: conditions — Schizophrenia; Motor Activity | interventions — Exercise; Cognitive Training; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized parallel assignment: Cognitive Training, Aerobic Exercise & Treatment as usual.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients are trained to not comment about the type of treatment they have been assigned to with the investigator who performs the assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise (Experimental): This program consists of an exercise dosage of 180 min/week administered in 3 sessions of 60 minutes. Each session includes 10 minutes of warm-up exercise before the main exercise and 10 minutes of cool-down afterwards.the principal exercise section includes 20 minutes of aerobic exercise and 20 minutes of resistance and strength exercises. The exercise intensity will be regulated according to the heart rate measured by a pulsimeter throughout the exercise. The target intensity level will be individualized according to the heart rate to set the moderate intensity level (HR values between ventilatory thresholds) and high intensity level (HR values from 2nd. ventilatory threshold to the peak threshold).
  Interventions: Behavioral: Aerobic Exercise
- Cognitive Training (Experimental): The CT group participates in a cognitive remediation program. This program consists of 3 sessions of 60 minutes per week. CT will be administered in groups of 5-8 subjects. The cognitive domains involved in the CT are attention/concentration, memory/learning, language, executive functions, social cognition, social skills, daily living activities and psychoeducation. Cognitive Remediation will be provided by using REHACOP, a cognitive remediation training tool designed and validated for Spanish patients with schizophrenia.
  Interventions: Behavioral: Cognitive Training
- Treatment as usual (Sham Comparator): The TaU Group receives the usual treatment that patients with schizophrenia in Spain enriched with occupational activities administered 3 times a week with a duration of 60 minutes each session.
  Interventions: Behavioral: Treatment as usual; Behavioral: Occupational Activities

INTERVENTIONS:
Behavioral: Aerobic Exercise — Physical exercise training consisting of aerobic exercise and strength/resistance training.
  Arms: Aerobic Exercise
Behavioral: Cognitive Training — Cognitive remediation program using REHACOP rehabilitation program.
  Arms: Cognitive Training
Behavioral: Treatment as usual — Standard care for schizophrenia + Leisure and free time activities.
  Arms: Treatment as usual
Behavioral: Occupational Activities — Engagement in activities aimed to keep patients actively involved in demanding tasks.
  Arms: Treatment as usual

SUMMARY:
This study evaluates the brain correlates of Cognitive Training and Aerobic Exercise in schizophrenia. A third of participants will receive Cognitive Training plus Standard Care for schizophrenia. Another third of participants will receive Aerobic Exercise Training plus Standard Care for schizophrenia. A control group will of participants will receive Standard Care plus Occupational Activities for the same duration and frequency as the experimental groups.

DETAILED DESCRIPTION:
This study, randomized, open, controlled with schizophrenia-standard-care, is aimed to determine structural and functional brain changes associated to cognitive remediation and physical exercise in schizophrenia.

The study participants will be enrolled in the catchment area of the Hospital Psiquiatrico de Alava, in the province of Alava, Basque Region, Northern Spain.147 patients diagnosed with schizophrenia will be randomly assigned to Cognitive Training Group or Aerobic Exercise Group or a Control Group for a five-month period.

Both Cognitive Training Group patients and Aerobic Exercise Group patients will participate in training sessions of 60 min/d, 3 d/wk. Patients assigned to Control Group will receive the standard care for schizophrenia in this area plus occupational activities for the same duration and frequency than the two experimental groups.

Cognitive Training will be implemented through REHACOP, a cognitive remediation program for Spanish speaking patients with schizophrenia whose efficacy on cognitive performance and negative symptoms has already been demonstrated in patients with schizophrenia. REHACOP is a "paper & pencil" based cognitive remediation program that covers 8 cognitive domains including social cognition. It is based on the principles of Optimization, Restauration & Compensation.

Aerobic Exercise Training will consist of an intensive physical exercise program supervised by certified graduates and doctorate students of Physical Activity and Sport Sciences. Sessions will include 10-minute warming-up and 10-minute back exercises and stretches. The main part of the session will consist of aerobic exercise (20-minute indoor bicycle) and muscle-resistance and strength exercises for 20 minutes. The intensity of the sessions will be determined on a case by case basis according to the HR necessary to achieve the intensity ranges (R2-moderate and R3-high). During the sessions, the bicycle's power and pace will be individually adjusted to achieve the selected HR.

The assessment batteries, neuroimaging and Serum BDNF levels will be administered and determined at baseline and immediately following the completion of the Cognitive Remediation or Aerobic Exercise interventions.

Primary outcomes: Structural and functional brain changes will be assessed by MRI neuroimaging. A Philips Achieva 3.0T MRI system equipped with a modular 32-channel architecture. 3 different types of images will be acquired: a) T1-weighted MRI imaging, b) Diffusion Tensor imaging, c) fMRI imaging at rest and using a cognitive paradigm.

Secondary outcomes will be changes in cognitive performance, clinical and functional changes and Serum BDNF changes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia (DSM-5 F20.9)
* More than 2 years since the onset of the disease.
* Stable cognitive impairment.
* Moderate severity of cognitive impairment in MATRICS scores (T score < 40 in, at least, 1 out of 7 cognitive domains).

Exclusion Criteria:

* Subjects clinically unstable (PANSS positive score > 19).
* Cognitive impairment due to another medical condition (neurocognitive disorders, brain injury, intellectual disability, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Grey Matter Volume Change | 5 months
  Assessment of Grey Matter volume changes (T1-weighted MRI) among the 3 groups using Voxel Based Morphometry (VBM).
Fractional Anisotropy Change | 5 months
  Assessment of changes in fractional anisotropy of White Matter fibers by Diffusion Tensor MR Imaging and using the Tract-Based Spatial Statistics (TBSS).
Functional Magnetic Resonance Imaging (fMRI) Change at Rest | 5 months
  Assessment of changes in fMRI at rest with the Coon Functional Connectivity Toolbox.
Functional Magnetic Resonance Imaging (fMRI) Change during the performance of a cognitive paradigm. | 5 months
  Assessment of changes in fMRI during the performance of a cognitive paradigm with Statistical Parametric Mapping (SPM8).

SECONDARY OUTCOMES:
Serum BDNF | 5 months.
  Assessment of changes in serum BDNF using ELISA immuno-assay techniques. Measured in ng/ml.
Clinical Symptoms of Schizophrenia measured by the Positive and Negative Symptoms Scale (PANSS). | 5 months.
  Severity of the negative symptoms will be assessed with the total score of the Subscale for Negative Symptoms of the PANSS scale, which comprises 7 items, each one measuring a specific negative symptom. Each item ranges from 1 (absence of the symptom) to 7 (extreme severity of the symptom). Total score of the Negative Subscale of the PANSS ranges from 7 (minimum score) to 49 (maximum severity). Severity of positive symptoms will be assessed with the total score of the Subscale for Positive Symptoms of the PANSS, which comprises 7 items ranging from 1 (absence of the symptom) to 7 (extreme severity of the symptom). Total score of the Positive Subscale ranges from 7 (minimun score) to 49 (maximun severity). General Psychopathology will be assessed with the total score of the General Psychopathology Subscale which comprises 16 items ranging from 1(absence of the symptom) to 7 (extreme severity of the symptom).
Negative Symptoms of Schizophrenia measured by the Brief Negative Symptoms Scale (BNSS). | 5 months
  Severity of negative symptoms will be assessed with the total score of the BNSS. Values ranges from 0 (total absence of negative symptoms) to 90 (maximum severity of negative symptoms).
Negative Symptoms of Schizophrenia measured by the Clinical Assessment Interview for Negative Symptoms Scale (CAINS) | 5 months
  Severity of negative symptoms will be assessed with the total score of the CAINS scale. Values ranges from 0 (total absence of negative symptoms) to 52 (maximum severity of negative symptoms).
Functional Outcome measured by the UCSD Performance Based Assessment of Functional Skills in Severe Mental Illness (UPSA). | 5 months
  The UPSA includes the following 5 subscales: Financial Skills, Communication, Comprehension/Planning, Transportation, Household Management. Total scores for each subscale are calculated by transforming raw scores into a 0- to-10 scale, yielding comparable scores on each scale. In order to have a 100-point summary score, each subscale score is multiplied by 2, yielding subscale scores ranging from 1 to 20. A summary UPSA score is calculated by summing these five scores, resulting in total scores ranging from 0 to 100. Scores of 0 represent maximum severity of functional impairment and a score of 100 represents total absence of functional disability.
Functional Outcome measured by the World Health Organization Disability Assessment Schedule (WHODAS 2.0). | 5 months
  The 36-item version of WHODAS 2.0 allows users to generate scores for the six domains of functioning and to calculate an overall functioning score. The scores assigned to each of the items - "none" (1), "mild" (2) "moderate" (3), "se- vere" (4) and "extreme" (5) - are summed. A score of 36 represents total absence of disability and 180 maximum severity of disability.
Functional Outcome measured by the Short Form (36) Health Survey (SF-36). | 5 months
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Physical Condition measured by the Modified Shuttle Walking Test | 5 months
  Heart rate achieved when walking between 2 cones spaced 10 meters at an increasing rate.
Cardiorespiratory Fitness measured with the Peak Oxygen Uptake (VO2 max) | 5 months
  maximum rate of oxygen consumption measured during incremental exercise (exercise of increasing intensity)
Weight. | 5 months
  Weight in Kg
Height | 5 months
  Height in meters.
Body composition measured with Body Mass Index (BMI) | 5 months.
  The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
Abdominal Perimeter | 5 months
  Abdominal perimeter measured in centimeters.
Body Composition measured with Total Body Water. | 5 months
  Percentage of Total Body Water measured by Bioimpedance.
Body Composition measured with Body Fat. | 5 months
  Percentage of Body Fat measured by Bioimpedance.
Blood Pressure (systolic and diastolic) | 5 months
  Blood Pressure (systolic and diastolic) measured in millimeters of mercury (mmHg)
Fasting Blood Glucose Levels | 5 months
  Fasting Blood Glucose Levels measured in mg/dl.
Fasting Cholesterol Levels | 5 months
  Fasting Cholesterol Levels measured in mg/dl.
Daily Physical Activity and Sedentary Behavior measured by the International Physical Activity Questionnaire. | 5 months
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.
Level of Daytime Sleepiness measured by Epworth Sleepiness Scale (ESS)ESS-EPWORTH. | 5 months
  The ESS measures a person's general level of daytime sleepiness, or their average sleep propensity in daily life (ASP). The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Intensity of Daily Physical Activity measured by the Accelerometer. | 5 months
  Measurement of body movement in terms of accelerations.
Cognition-Processing Speed | 5 months
  WAIS III test: Digit Symbol-Coding. Measured in number of symbols correctly entered in 2 minutes.
Cognition-Attention/Vigilance Stroop Test | 5 months
  Stroop Test: measured in the number of items read or named in 45 seconds for each of the three sheets (word, color, and color-word).
Cognition-Working Memory Digit Span Backward | 5 months
  WAIS IV test: Digit Span Backward subtest. Measured with the number of sequences of numbers recalled in inverse order.
Cognition-Verbal Learning/Memory | 5 months
  Hopkins Verbal Learning Test-Revised (HVLT-R): number of correct words recalled.
Cognition-Reasoning/Problem Solving | 5 months
  Modified Wisconsin Card Sorting Test (M-WCST): score achieved at the M-WCST.
Cognition-Cognitive Reserve | 5 months
  Spanish version of the Word Accentuation Test (TAP-E). Measured with the number of correct attempts.
Cognition-Figural Creativity | 5 months
  Torrance Test of Creative Thinking: Picture Completion subtest. Measured with Fluency, Originality, Elaboration, Resistance to Premature Closure, Abstractness of Titles, and Creative Strengths dimensions obtained from the drawings made in the task.
Cognition-Verbal Creativity | 5 months
  Torrance Test of Creative Thinking: Unusual Uses subtest. Measured with Fluency, Originality, and Flexibility dimensions obtained from the written unusual uses for cardboard boxes and tin cans.
Social Cognition-Social Attribution | 5 months
  Social Attribution Test (SAT). SAT is comprised of a 64 second animation with geometric figures enacting a social drama and 19 multiple-choice questions about the animation. Four possible responses are given to each question. Each correct response is scored with 1 point. Total score ranges from 0 to 19.
Social Cognition-Emotion Recognition | 5 months
  Bell Lysaker Emotion Recognition Task (BLERT). BLERT consists of 21 short video clips in which an actor displays one of seven emotions with three neutral monologues. The examinee is asked to indicate which emotion the actor is portraying. Each correct response is scored with 1 point. The total score is obtained from the sum of each correct emotion recognition, ranging from 0 to 21.
Social Cognition-Theory of Mind | 5 months
  Happe's "Strange Stories Task" Test. Strange Stories Task is comprised of 8 stories concerning double bluff, mistakes, persuasion, and white lies. Each story is scored from 0 to 2. Higher scores indicate a better performance in theory of mind.
Social Functioning measured by the Social Functioning Scale Short-Form (SFS-15) | 5 months
  The SFS-15 is a 15-item scale designed to measure social functioning in patients with schizophrenia. It includes items about isolation, interpersonal communication, independence-execution, independence-competence, and employment-occupation. 13 of the items range from 0 to 3 and the other 2 items range from 1 to 2. Total score is obtained from the sum of the 15 items. Total score range from 1 to 43 points. Higher scores indicate higher level of social functioning.
Self-Efficacy measured by the General Self-Efficacy Scale | 5 months
  General Self-Efficacy Scale is a 10-item scale that measures optimistic self-beliefs to cope with a variety of difficult demands in life. The scores assigned to each of the item - "Not at all true" (1), "Hardly true" (2), "Moderately true" (3), and "Exactly true" (4) - are summed. The final score ranges from 10 to 40, higher scores indicating a higher level of self-efficacy.
Social Anhedonia measured with the Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) | 5 months
  The ACIPS is a 17-item scale that consists of 7 anticipatory and 10 consummatory items. The scores assigned to each of the items range from 1 (very false for me) to 6 (very true for me). Total score is obtained from the sum of the 17 items. Higher scores indicate higher ability to experience interpersonal pleasure.
Handedness measured by the Edinburgh Handedness Inventory | 5 months
  A self-report questionnaire assessing the dominance of a person's right or left hand in ten different everyday activities.
Treatment satisfaction measured by the Spanish version of Consumer Reports Effectiveness Scale (CRES-4) | 5 months
  CRES-4 consists of a 4-item scale designed to evaluate patient's satisfaction with the received therapy. Its global score reflects treatment effectiveness as perceived by the patient. 3 components can be obtained: "satisfaction" (based on the first item, which ranges from 0 to 5), "problem resolution" (based on the second item, which ranges from 0 to 5), and "perceived emotional change" (obtained from the subtraction of the third from the fourth item, which range from 0 to 4). The "satisfaction" component is multiplied by 20, the "problem resolution" by 20 and the "perceived emotional change" by 12.5. Final score is obtained from the sum of the three components, ranging from 0 to 300. Higher scores indicate a greater perception of treatment efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro M Sanchez Gomez, MD, Principal Investigator — Hospital Psiquiatrico de Alava. Red de Salud Mental de Araba.
Locations (1):
- Hospital Psiquiatrico de Alava. Red Salud Mental de Araba, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sanchez P, Pena J, Bengoetxea E, Ojeda N, Elizagarate E, Ezcurra J, Gutierrez M. Improvements in negative symptoms and functional outcome after a new generation cognitive remediation program: a randomized controlled trial. Schizophr Bull. 2014 May;40(3):707-15. doi: 10.1093/schbul/sbt057. Epub 2013 May 18. PMID 23686130
- [Result] Ojeda N, Pena J, Bengoetxea E, Garcia A, Sanchez P, Elizagarate E, Segarra R, Ezcurra J, Gutierrez-Fraile M, Eguiluz JI. [REHACOP: a cognitive rehabilitation programme in psychosis]. Rev Neurol. 2012 Mar 16;54(6):337-42. Spanish. PMID 22403146
- [Result] Pena J, Ibarretxe-Bilbao N, Sanchez P, Uriarte JJ, Elizagarate E, Gutierrez M, Ojeda N. Mechanisms of functional improvement through cognitive rehabilitation in schizophrenia. J Psychiatr Res. 2018 Jun;101:21-27. doi: 10.1016/j.jpsychires.2018.03.002. Epub 2018 Mar 6. PMID 29525739
- [Result] Pena J, Ibarretxe-Bilbao N, Sanchez P, Iriarte MB, Elizagarate E, Garay MA, Gutierrez M, Iribarren A, Ojeda N. Combining social cognitive treatment, cognitive remediation, and functional skills training in schizophrenia: a randomized controlled trial. NPJ Schizophr. 2016 Nov 9;2:16037. doi: 10.1038/npjschz.2016.37. eCollection 2016. PMID 27868083
- [Result] Ojeda N, Pena J, Bengoetxea E, Garcia A, Sanchez P, Elizagarate E, Segarra R, Ezcurra J, Gutierrez-Fraile M, Eguiluz JI. [Evidence of the effectiveness of cognitive rehabilitation in psychosis and schizophrenia with the REHACOP programme]. Rev Neurol. 2012 May 16;54(10):577-86. Spanish. PMID 22573504
- [Result] Ojeda N, Pena J, Sanchez P, Bengoetxea E, Elizagarate E, Ezcurra J, Gutierrez Fraile M. Efficiency of cognitive rehabilitation with REHACOP in chronic treatment resistant Hispanic patients. NeuroRehabilitation. 2012;30(1):65-74. doi: 10.3233/NRE-2011-0728. PMID 22349843
- [Derived] Tous-Espelosin M, Pavon C, Elizagarate E, Sampedro A, Maldonado-Martin S. As We Were and As We Should Be, Combined Exercise Training in Adults With Schizophrenia: CORTEX-SP Study Part II. Scand J Med Sci Sports. 2024 Aug;34(8):e14707. doi: 10.1111/sms.14707. PMID 39054763
- [Derived] Tous-Espelosin M, de Azua SR, Iriarte-Yoller N, MartinezAguirre-Betolaza A, Sanchez PM, Corres P, Arratibel-Imaz I, Sampedro A, Pena J, Maldonado-Martin S. Clinical, physical, physiological, and cardiovascular risk patterns of adults with schizophrenia: CORTEX-SP study: Characterization of adults with schizophrenia. Psychiatry Res. 2021 Jan;295:113580. doi: 10.1016/j.psychres.2020.113580. Epub 2020 Nov 18. PMID 33246589